CLINICAL TRIAL: NCT01601782
Title: Impact of Volume Imaging With Ultrasound
Brief Title: Impact of Volume Imaging Using Diagnostic Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was determined that the volume imaging was not working.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jon Jacobson, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00030780
Record Dates: First submitted 2012-05-01; First posted 2012-05-18 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Bone Injuries; Muscle Injuries; Tendon Injuries
MeSH Terms: conditions — Tendon Injuries | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volume Imaging scan (Experimental): New type of ultrasound scan using General Electric US scanner, Model is a GE Logiq E9.
  Interventions: Procedure: Ultrasound Scan; Device: Ultrasound Scan using a General Electric Ultrasound Scanner Model Logiq E9 (model name).

INTERVENTIONS:
Procedure: Ultrasound Scan — Subject will be required to lie flat for no longer than 3 minutes to complete a volume imaging ultrasound scan of the injured area. Following the volume imaging scan a conventional ultrasound scan will be completed as ordered by their clinician.
  Other Names: Volumetric Ultrasound; 3D Ultrasound Imaging; Volume Imaging
Device: Ultrasound Scan using a General Electric Ultrasound Scanner Model Logiq E9 (model name). — The subject will be required to lie flat for approximately 5 to 10 minutes to complete a conventional ultrasound scan to x-ray the muscle and tendon injuries.

SUMMARY:
Determine if volume imaging can diagnose bone, ligament, muscle injuries.

DETAILED DESCRIPTION:
The investigators are attempting to determine if Volume imaging (a new type of ultrasound imaging)can accurately diagnose injuries of the muscle ligaments, tendons and bones when compared to conventional ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Must be scheduled to have a musculoskeletal (bone, ligament, muscle, tendon) ultrasound performed as part of their routine clinical care.

Exclusion Criteria:

* Unable to lie flat on ultrasound table.
* Subjects under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Jacobson, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who are referred for an ultrasound of the extremity will be asked to participate in the study.
Groups:
- Volume Imaging Scan: New type of ultrasound scan using General Electric US scanner, Model is a GE Logiq E9.
  Ultrasound Scan using a General Electric Ultrasound Scanner Model Logiq E9 (model name). : The subject will be required to lie flat for approximately 5 to 10 minutes to complete a conventional ultrasound scan to image the muscle and tendon injuries.
  Ultrasound Scan : Subject will be required to lie flat for no longer than 3 minutes to complete a volume imaging ultrasound scan of the injured area. Following the volume imaging scan a conventional ultrasound scan will be completed as ordered by their clinician.
Period: Overall Study
Arm/Group | Volume Imaging Scan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients were randomly evaluated without pre-selection of gender or race
Arm/Group | Volume Imaging Scan
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 25 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of 3D Ultrasound Scanning Expressed as Percent Correlation Between Images From Conventional Ultrasound and Volume Imaging
Description: Both ultrasound and volume imaging scans were done on the same day. For all scanned patients, the ultrasound technologist took a volume of images focusing where the patient had symptoms. The study PI reviewed the images, then went back in to do second scan. It took 5 to 10 minutes to complete a conventional ultrasound scan and up to 3 minutes to complete a volume imaging ultrasound scan.
Time Frame: Up to 13 minutes
Measure: Number; unit: percent correlation
Arm/Group | Volume Imaging Scan
Number analyzed (Participants) | 16
percent correlation | NA — Two sets of images were collected for all 16 participants. In each case the volume imaging was not sufficiently clear to allow for the diagnostic interpretation necessary to support any numerical correlation between the two scans.

ADVERSE EVENTS:
Time Frame: up to 1 hour
Arm/Group | Volume Imaging Scan
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
16 patients were studied as part of a pilot project to determine if 3D ultrasound offers any benefit over routine standard ultrasound imaging of the extremity. The study was terminated after evaluating 16 subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No